CLINICAL TRIAL: NCT05704829
Title: NeoAdjuvant Dynamic Marker - Adjusted Personalized Therapy Comparing Trastuzumab-deruxtecan Versus Pacli-/Docetaxel+Carboplatin+Trastuzumab+Pertuzumab in HER2+ Early Breast Cancer
Brief Title: NeoAdjuvant Therapy With Trastuzumab-deruxtecan Versus Chemotherapy+Trastuzumab+Pertuzumab in HER2+ Early Breast Cancer
Acronym: ADAPTHER2-IV
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM12 (ADAPT-HER2-IV)
Record Dates: First submitted 2022-12-28; First posted 2023-01-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Early Breast Cancer
Keywords: HER2+; T-DXd; Trastuzumab-deruxtecan; pCR; intermediate risk; high risk; low risk; recurrence; neoadjuvant
MeSH Terms: conditions — Recurrence | interventions — trastuzumab deruxtecan; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multicentre, interventional, prospective, two-arm, randomised, open-label, controlled (neo-)adjuvant, phase-II trial evaluating the efficacy and safety of trastuzumab-deruxtecan (T-DXd) vs. standard-of-care paclitaxel + trastuzumab + pertuzumab (PAC+T+P) in low- to intermediate-risk or docetaxel/paclitaxel + carboplatin + trastuzumab + pertuzumab in intermediate- to high-risk HER2+ early breast cancer in pre- and postmenopausal women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T-DXd: HER2+ and low-intermediate risk for recurrence (Experimental): 12 weeks T-DXd i.v. in neoadjuvant treatment; pCR dependent T-DXd for 1 year in total in postneoadjuvant treatment
  Interventions: Drug: Trastuzumab deruxtecan
- T-DXd: HER2+ and intermediate-high risk for recurrence (Experimental): 18 weeks T-DXd i.v. in neoadjuvant treatment; pCR dependent T-DXd for 1 year in total in postneoadjuvant treatment
  Interventions: Drug: Trastuzumab deruxtecan
- Control: HER2+ and low-intermediate risk for recurrence (Other): Standard-of-Care-Treatment: 12 weeks PAC+T+P (standard-of-care) in neoadjuvant treatment; pCR dependent SOC chemotherapy +T+/-P or SOC T+/-P for 1 year in total in postneoadjuvant treatment
  Interventions: Drug: Standard-of-Care
- Control: HER2+ and intermediate-high risk for recurrence (Other): Standard-of-Care-Treatment: 18 weeks PAC/DOC+Carbo+T+P (standard-of-care) in neoadjuvant treatment; pCR dependent SOC chemotherapy +T+/-P or SOC T+/-P for 1 year in total in postneoadjuvant treatment
  Interventions: Drug: Standard-of-Care

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — T-DXd i.v.
  Other Names: ENHERTU
  Arms: T-DXd: HER2+ and intermediate-high risk for recurrence; T-DXd: HER2+ and low-intermediate risk for recurrence
Drug: Standard-of-Care — Chemotherapy+T+P
  Other Names: Chemotherapy+T+P
  Arms: Control: HER2+ and intermediate-high risk for recurrence; Control: HER2+ and low-intermediate risk for recurrence

SUMMARY:
ADAPT-HER2-IV will address question of optimal neoadjuvant therapy in patients with less advanced -HER2+ EBC.

ADAPT-HER2-IV is planned as a superiority trial to demonstrate higher pCR rates in both clinically relevant subgroups of low-intermediate risk HER2+ EBC. Moreover, it aims to demonstrate excellent survival in patients treated by T-DXd (with the use of standard chemotherapy at investigator´s decision restricted only to patients with substantial residual tumour burden after T-DXd-treatment).

DETAILED DESCRIPTION:
As the ADAPT-trials have clearly shown, pCR after 12 weeks of therapy, independent of the specific de-escalated neoadjuvant regimen and independent of further use of systemic chemotherapy, is an independent predictor of excellent prognosis4,19, also in patients treated by an antibody-drug conjugate alone (T-DM1), or in those receiving pertuzumab+trastuzumab+/-weekly paclitaxel.

In contrast to the adjuvant setting, none of the neoadjuvant trials so far has focused on HER2+ patients with a low-intermediate risk profile (e.g., node-negative patients with cT1-2 tumours). The ADAPT-HER2-IV trial aims to close this evidence gap.

Since there is some uncertainty about the optimal treatment duration in intermediate- to high-risk HER2+ EBC (e.g., tumour size >3 cm), we recommend using a longer 18-week taxane-based treatment (+/- carboplatin, at investigator´s decision) due to a large body of evidence for taxane + carboplatin combinations in patients in locally advanced stages.

Antibody-drug conjugates appear to be ideal candidate drugs for a "de-escalated" treatment due to their favourable safety (reduced alopecia, polyneuropathy rates, etc.) and a high efficacy profile (e.g., comparable pCR rates after 18 weeks of T-DM1 and taxane+pertuzumab+trastuzumab in the PREDIX HER2 trial20). Similarly to the classical chemotherapy landscape, optimal duration of antibody-drug conjugate-based neoadjuvant therapy remains unclear. pCR rates of around 40% to 60% were observed after 12 and 18 weeks of T-DM1 treatment (+/-pertuzumab) in the ADAPT TP, KRISTINE and PREDIX HER2 trials in HR+/HER2+ disease21,22. Moreover, long-term survival seem to be comparable between T-DM1+pertuzumab and older chemotherapy-containing regimens (docetaxel+carboplatin+trastuzumab+pertuzumab) despite of higher local progression rates and lower pCR in one study22.

Trastuzumab-deruxtecan (T-DXd) has shown promising activity in a small cohort of metastatic patients, including both HER2+ and HER2-low BC, pre-treated with several lines of therapy. Doi et al. reported overall response rates (ORR) of 58% and a disease control rate of 100% with overall survival at 12 months at in HER2+ disease pre-treated by T-DM1+/-pertuzumab in a late line setting23. T-DXd-therapy was associated with a manageable safety profile. Recently, clearly higher efficacy of T-DXd vs. T-DM1 was shown in second line metastatic breast cancer (MBC) in the DESTINY-03 trial24. Median progression free survival was not reached in T-DM1-arm vs. 6.8 months in the T-DXd-arm. This effect was independent of hormone receptor status, prior pertuzumab treatment, visceral metastases, number of prior therapy lines and presence of brain metastases. ORR was doubled (34.2 vs. 79.7%), favouring the T-DXd arm.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet all the following criteria:

1. Female patients with invasive, untreated HER2+ breast cancer (as assessed by local pathology) maximum 6 weeks before registration (standard-of-care diagnostic biopsy according to current AGO guidelines)
2. Age ≥18 years 3a. Cohort 1: low- to intermediate-risk for recurrence as per investigator´s decision (recommendation: cT1c - cT2 (1 - ≤3cm), cN0; cT1a/b excluded), OR 3b. Cohort 2: intermediate- to high-risk for recurrence as per investigator´s decision (recommendation: cT2 (>3 - ≤5cm), cN0) 3c. Elderly patients (≥ 65 years) may be assigned to any cohort as per investigator's decision

4. Written informed consent 5. LVEF ≥ 50% within 28 days before randomisation 6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1 7. Adequate organ and bone marrow function within 14 days before randomisation 8. Adequate treatment washout period before randomisation (refer to protocol for detailed information) 9. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential (refer to protocol for detailed information) 10. Female subjects must not donate, or retrieve for their own use, ova from the time of randomisation and throughout the study treatment period, and for at least 7 months after the final study drug administration. (refer to protocol for detailed information)

Exclusion Criteria:

Patients eligible for inclusion in this study must not meet any of the following criteria:

1. Non-operable breast cancer including inflammatory breast cancer
2. cT1a/b breast cancer
3. Any previous history of invasive breast cancer
4. Primary malignancies within 5 years, with the exception of adequately resected non-melanoma skin cancer, curatively treated in-situ disease
5. Any evidence for existing metastatic disease (confirmed by CT Thorax/Abdomen, bone scan, or other methods according to clinical practice
6. Previous or concurrent treatment with cytotoxic agents for any reason (except non-oncological reasons)
7. Concurrent treatment with other experimental drugs and participation in another clinical trial with any investigational drug within 30 days prior to study entry
8. Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study/inadequate organ function
9. Reasons indicating risk of poor compliance
10. Woman of child-bearing potential defined as a woman physiologically capable of becoming pregnant, and not using highly effective methods of contraception during the study treatment and for 3 months after stopping the treatment.
11. Use of oral (oestrogen and progesterone), transdermal, injected, or implanted hormonal methods of contraception as well as hormonal replacement therapy.
12. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
13. Patients with a medical history of myocardial infarction (MI) within 6 months before randomisation, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrolment to rule out MI.
14. Corrected QT interval (QTcF) prolongation to > 470 msec (females) based on average of the screening triplicate12-lead ECG.
15. History of (non-infectious) ILD / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
16. Lung criteria: Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder; Any autoimmune, connective tissue or inflammatory disorders (e.g., Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of randomisation; Prior pneumonectomy (complete); Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
17. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients should be tested for HIV prior to randomisation if required by local regulations or ethics committee (EC).
18. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan.

    Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IMP.
19. Known allergy or hypersensitivity to study treatment (T-DXd) or any of the study drug excipients.
20. History of severe hypersensitivity reactions to other monoclonal antibodies.
21. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
1. pCR rate after neoadjuvant treatment | after 12 weeks of neoadjuvant treatment
  defined as ypT0is/ypN0, to be compared between all T-DXd treated patients versus standard-of-care (PAC+T+P or PAC/DOC+Carbo+T+P) (pooled across cohorts)
1. pCR rate after neoadjuvant treatment | after 18 weeks of neoadjuvant treatment
  defined as ypT0is/ypN0, to be compared between all T-DXd treated patients versus standard-of-care (PAC+T+P or PAC/DOC+Carbo+T+P) (pooled across cohorts)
2. distant disease-free survival (dDFS, according to STEEP 2.0 criteria) | after 3 years
  distant disease-free survival (dDFS, according to STEEP 2.0 criteria) in T-DXd treated patients (pooled across cohorts)

SECONDARY OUTCOMES:
clinical response | after 6 weeks of treatment
  clinical response after 6 weeks of treatment
clinical response | after 12 weeks of treatment
  clinical response after 12 weeks of treatment
clinical response | after 18 (cohort 2) weeks of treatment
  clinical response after 18 (cohort 2) weeks of treatment
dDFS in patients with pCR | after 3 years
  dDFS in patients with pCR after neoadjuvant treatment without further chemotherapy
pCR rates after different treatment durations | 12 versus 18 weeks
  Comparison of pCR rates after different treatment durations (12 versus 18 weeks) of both treatments in pooled cohorts
pCR rates in T-DXd 12 weeks versus PAC+T+P | after 12 weeks
  Comparison of pCR rates in T-DXd 12 weeks versus PAC+T+P
pCR rates in T-DXd 18 weeks versus PAC/DOC+Carbo+T+P | after 18 weeks
  Comparison of pCR rates in T-DXd18 weeks versus PAC/DOC+Carbo+T+P
iDFS | at end of study
  survival endpoint STEEP 2.0
OS | at end of study
  survival endpoint STEEP 2.0
LRFS | at end of study
  survival endpoint STEEP 2.0
BCFS | at end of study
  survival endpoint STEEP 2.0
DRFI | at end of study
  survival endpoint STEEP 2.0
QOL | after 1 year
  health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Centre, Dept. Obstetrics & Gynaecology and CCC Munich LMU University Hospital; Sherko Kuemmel, PRof. Dr., Principal Investigator — Breast Centre, Kliniken Essen Mitte Essen; Oleg Gluz, PD Dr., Principal Investigator — Breast Centre, Evang. Bethesda-Hospital Moenchengladbach; Michael Braun, Prof. Dr., Principal Investigator — Breast Centre Rotkreuzklinikum Munich; Monika Graeser, PD Dr., Principal Investigator — Breast Centre, Evang. Bethesda-Hospital Moenchengladbach
Locations (43):
- Germany (43):
  - Klinikum Mittelbaden, Brustzentrum, Baden-Baden, Baden-Wurttemberg
  - Praxis für Interdisziplinäre Onkologie und Hämatologie (PIO), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Hämotologisch onkologische Praxis Heinrich Bangerter Augsburg GbR, Augsburg, Bavaria
  - Universitätsklinikum Augsburg / Klinik für Frauenheilkunde und Geburtshilfe, Augsburg, Bavaria
  - Breast Center of the University of Munich (LMU) Universitätsfrauenklinik, Munich, Bavaria
  - Rotkreuz Klinikum München, Munich, Bavaria
  - Klinikum Bremerhaven Reinkenheide, Bremerhaven, City state Bremen
  - Universittsklinikum am Klinikum Südstadt, Rostock, ecklenburg-Vorpommerns
  - AGAPLESION Markus Krankenhaus Gynäkologie, Frankfurt am Main, Hesse
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main, Hesse
  - Klinikum Kassel, Kassel, Hesse
  - Studien GbR Braunschweig, Braunschweig, Lower Saxony
  - Niels-Stensen-Kliniken Franziskus-Hospital, Georgsmarienhütte, Lower Saxony
  - Ärztehaus am Bahnhofsplatz, Hildesheim, Lower Saxony
  - MVZ Klinik Dr. Hancken GmbH, Stade, Lower Saxony
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld, North Rhine-Westphalia
  - St. Elisabeth Krankenhaus GmbH, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln GmbH / Brustzentrum Holweide, Cologne, North Rhine-Westphalia
  - Kliniken für Frauenheilkunde / Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Luisenkrankenhaus GmbH, Düsseldorf, North Rhine-Westphalia
  - Sankt-Antonius-Hospital, Eschweiler, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Klinik für Senologie/Interdisziplinäres Brustzentrum, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Brustzentrum, Essen, North Rhine-Westphalia
  - Onkodok Gütersloh, Gütersloh, North Rhine-Westphalia
  - St. Barbara Klinik, Hamm, North Rhine-Westphalia
  - Brustzentrum Niederrhein, Johanniter Bethesda Krankenhaus, Mönchengladbach, North Rhine-Westphalia
  - MVZ Media Vita am St. Franziskus Hospital, Münster, North Rhine-Westphalia
  - Frauenklinik St. Louise-St. Vincenz-KH GmbH, Paderborn, North Rhine-Westphalia
  - MKS St. Paulus GmbH, Schwerte, North Rhine-Westphalia
  - Praxisnetzwerk Hämatologie und intern. Onkologie, Troisdorf, North Rhine-Westphalia
  - Helios-Klinik Wuppertal, Wuppertal, North Rhine-Westphalia
  - Klinikum Mutterhaus, Trier, Rhineland-Palatinate
  - CaritasKlinikum Saarbrücken St. Theresia, Saarbrücken, Saarland
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Frauenklinik / Brustzentrum am Klinikum Obergölzsch Rodewisch, Rodewisch, Saxony
  - UK Schleswig Holstein, Lübeck, Schleswig-Holsteins
  - Charite Campus Mitte, Berlin
  - Ev. Waldkrankenhaus Spandau, Berlin
  - Universitätsklinikum Hamburg-Eppendorf / Klinik und Poliklinik für Gynäkologie, Hamburg
  - Brustzentrum am Krankenhaus Jerusalem, Hamburg

IPD SHARING:
Plan to Share IPD: No